CLINICAL TRIAL: NCT03829202
Title: Comparison of Gait and Functional Performance Between RheoKnee and Mechanical Knee in K2 and K3 Users: A Single-Subject Design
Brief Title: Evaluation of Transfemoral Amputees When Transitioning From a Mechanical to a Microprocessor Prosthetic Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Methodist Rehabilitation Center (Other)
Collaborators: Össur Iceland ehf (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MRC_Ossur_MPK
Record Dates: First submitted 2019-01-16; First posted 2019-02-04 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Amputation of Lower Limb Above Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A-B-A Group (Experimental): Daily use of own mechanical knee for 4 weeks (A), followed by RheoKnee microprocessor prosthetic knee for 4 weeks (B), and concluding with own mechanical knee for 4 weeks (A).
  Interventions: Device: Own mechanical knee; Device: RheoKnee microprocessor prosthetic knee
- B-A-B Group (Experimental): Daily use of RheoKnee microprocessor prosthetic knee for 4 weeks (B), followed by own mechanical knee for 4 weeks (A), and concluding with RheoKnee microprocessor prosthetic knee for 4 weeks (B).
  Interventions: Device: Own mechanical knee; Device: RheoKnee microprocessor prosthetic knee

INTERVENTIONS:
Device: Own mechanical knee — Daily use of own mechanical knee
Device: RheoKnee microprocessor prosthetic knee — Daily use of RheoKnee microprocessor prosthetic knee
  Other Names: MPK

SUMMARY:
The central hypothesis of this proposal is that real-life benefits of microprocessor knees (MPK) are largely underappreciated because of the lack of sensitive and ecologically valid methods for evaluating motor performance. This makes it difficult to justify MPKs for many amputees who could benefit from it. Using recently developed outcome measures shown to be more effective in evaluating prosthesis users than commonly employed metrics, 7 transfemoral prosthesis users who exclusivity utilize a non-microprocessor mechanical knee were evaluated as they transitioned to and from an MPK in an ABA/BAB single subject design protocol. Subjects were also evaluated with existing clinical measures established for lower limb amputees.

DETAILED DESCRIPTION:
Research Hypothesis The central hypothesis of this proposal is that real-life benefits of microprocessor knees (MPK) are largely underappreciated because of the lack of sensitive and ecologically valid methods for evaluating motor performance. This makes it difficult to justify MPKs for many amputees who could benefit from it. The investigators' recent research on the stride length-cadence relationship and dual-task gait analysis offers a new direction to overcome some of these limitations.

Why stride length-cadence relationship for MPKs? Because stride length and cadence form a strong linear relationship over a range of gait velocities, examining the strength of their association offers a unique way to characterize natural gait. The investigators found that the stride length-cadence relationship is disrupted in prosthesis users. Also, the step length-cadence relationship is disrupted bilaterally, indicating altered neurocontrol of gait. Unlike a mechanical knee, MPKs adjust properties to accommodate changes in velocity, resembling more natural gait pattern. Thus, the stride length-cadence relationship is expected to be tighter for MPKs than a mechanical knee.

Why dual-task gait for MPKs? Dual-task gait is the act of walking while performing an additional task (talking, texting, etc.). The additional load imposed on the nervous system alters gait. Thus, "walking while talking" better reflects real-life gait than standard gait analysis. Dual-task gait studies in prosthetic users are rare. The classic outcome measure in dual-task studies is a standard deviation divided by the mean for each gait parameter separately, which ignores their dependence on changes in speed. The investigators recently developed a new method for analyzing dual-task gait based on the linear relationship that stride length and cadence have with velocity. The standard deviations of the difference between the actual data point for stride length or cadence from the point predicted by the line that represents the best fit with velocity are compared between the free walking and dual-task walking. This calculation of variability in stride length or cadence accounts for their trial-to-trial changes with the velocity that can influence results. Previous studies indicate that MPKs require less additional thought during gait. If indeed the case, the users should be able to shift motor and cognitive resources from gait to other activities and, at the same time, have less variable gait under dual-task condition. Since decreased gait variability has been related to better neurocontrol of gait and lesser risk for falls, the proposed proof-of-principle study will be the first step toward providing critical missing evidence for justifying the use of MPKs in a broader population of amputees, particularly in K2 users or persons with cognitive impairments as a result of vascular disease or diabetes.

Objective: Evaluate differences in gait and function between an MPK (RheoKnee®, Ossur) and a mechanical knee in K2 and K3 prosthesis users in an A-B-A and B-A-B single-subject design.

Specific Aim 1: Assess the stride length-cadence relationship during gait with the MPK compared to the mechanical knee.

Hypothesis 1.1: The stride length-cadence linear relationship will significantly improve after wearing the MPK. Hypothesis 1.2: The linearity of the stride length-cadence relationship will be significantly higher for the MPK than the mechanical knee.

Specific Aim 2: Determine the changes in dual-task cost while walking with the MPK compared to the mechanical knee.

Hypothesis 2.1: Under the dual-task condition, the variability in stride length and cadence will be significantly smaller while wearing the MPK than the mechanical knee.

Specific Aim 3: Compare the performance between the MPK and the mechanical knee on clinical measures of mobility, balance, and user preference.

Hypothesis 3.1: Measures of functional mobility will improve more while wearing the MPK than the mechanical knee Hypothesis 3.2: Balance measures will improve more while wearing the MPK more than the mechanical knee.

Hypothesis 3.3: Joint range of motion and ground reaction force symmetry will improve while wearing the MPK.

Study Design:

The study will use an A-B-A and B-A-B single-subject design (A- the subject's current mechanical knee; B- MPK: RheoKnee®). The purpose of B-A-B design is to control for a learning effect due to multiple repetitions of cognitive tasks during dual-task gait, which may contribute to hypothesized improvements in phase B of the A-B-A design. Each phase will last 4 weeks.

Protocol:

Eligible subjects who signed the consent form will be randomly allocated to the A-B-A or B-A-B group. The proper fit/alignment of the current mechanical knee will be verified, and, if fine, the 3D gait analysis and functional assessment (Full Evaluation) will be performed at baseline. Walking at up to 5 self-selected speeds (very slow to very fast) and dual-task gait (Gait Evaluation) will also be evaluated at baseline and then on a weekly basis throughout each phase. At the end of each phase, Gait Evaluation and Full Evaluation are repeated. The end of each current phase and the beginning of a new phase are separated by a transition period. The transition period starts with the alignment of a new device followed by 2 weeks of accommodation during which up to 6 gait training sessions are provided by a physical therapist (PT) and the alignment is checked. All efforts will be made to maintain the subject's current socket style and suspension system. The B-A-B design is identical to the A-B-A design except for an additional transition period at the very beginning since the naive subjects are fit for the first time with the MPK.

Methods:

Users of a mechanical prosthetic knee will be recruited from the population served by Methodist Rehabilitation Center if they meet the enrollment criteria. After signing the consent form, the subjects will be allocated to the A-B-A or B-A-B group using a random number sequence.

Gait Evaluation:

Self-Selected Speeds:

Temporal and spatial footfall data will be collected by an electronic walkway (20 ft) as the subject walks at five self-selected speeds (very slow, slow, normal, fast, very fast). An area at each end of the walkway will allow for acceleration and deceleration so that only steady-state gait is recorded. Subjects will complete a minimum of 4 passes at each speed, which they will freely select to achieve the most natural walking pattern. The normal gait speed will always be collected first. The order of slower/faster speed categories will be randomized with the very slow/fast speed collected last in each category. Subjects will be instructed to modulate the speed within safety limits and encouraged to complete all speeds, to the extent possible.

Dual-Task Gait:

Four cognitive tasks will be used for dual-task gait; backward spelling, serial subtraction, digit span, and category listing. Three tasks will be used at each assessment point to curb the effect of learning. Tasks will be selected at random so that each is given an equal number of times in each phase. All four tasks will be used at baseline. Different prompts will be given to ensure no task is presented the same way twice.

Before each assessment, the subject will practice the selected tasks while seated to familiarize with the protocol. For the dual-task gait, the subject will be instructed to walk at a comfortable pace and simultaneously perform cognitive tasks without specific instructions on prioritization. The cognitive tasks will be block randomized with each block containing 4 walking trials. At the end, the subject will be asked to rate the task difficulty on a 7-point Likert scale.

Full Evaluation:

* Functional prosthetic assessment (Amputee Mobility Predictor, L-test, 6-minute Walk Test, Berg Balance Scale, Physiological Cost Index,Temporal/Spatial Gait Assessment)
* User evaluation of the prosthesis (Prosthesis Evaluation Questionnaire, study specific knee preference evaluations)
* Computerized 3D gait assessment (3D gait kinematics and kinetics)
* Cognition/mood (Modified Mini-Mental State Exam, Trails A & B, Patient Health Questionnaire)

Outcome Measures:

Specific Aim 1: Stride-length cadence relationship

* Main outcome: coefficient of determination (R2) of the linear regression line
* Secondary outcomes: peak velocity & range of velocities

Specific Aim 2: Cost of dual-task gait

* Main outcome: variability (standard deviation) of stride length and cadence under unconstrained and dual-task conditions
* Secondary outcomes: peek/range of velocities under the two conditions; the rating of difficulty

Specific Aim 3: Comparison of change between K2 and K3 users

* Main outcomes: scores from the Berg Balance Scale, Prosthesis Evaluation Questionnaire, Amputee Mobility Predictor, L-test, 6-minute Walk Test, Physiological Cost Index
* Secondary outcomes: Temporal/Spatial Gait Assessment, 3D joint range of motion, joint angles at critical instants, the ground reaction force

Analysis:

Due to the nature of the single-subject design, the data will be evaluated both qualitatively and with small-n design statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral above-knee amputation
* Exclusive use of an non-microprocessor knee for more than 1 year
* Comfortable socket fit
* No skin breakdown on the residual limb
* Medicare functional classification level 2 or 3
* Ability to read or understand English
* Ability to walk 10 m with or without an assistive device

Exclusion Criteria:

* Cognitive or general health problems that would prevent participation in the study
* Physical limitations on the non amputated side

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-12-19 (Actual); Primary Completion 2014-08-12 (Actual); Study Completion 2014-08-12 (Actual)

PRIMARY OUTCOMES:
Stride Length-Cadence Relationship | Weekly for the duration of the study, approximately 15 weeks
  The stride length-cadence relationship measures the coordination between the temporal and spatial gait parameters over a range of walking speeds. Greater correlation represents improved gait coordination.
Dual-task residual standard deviation | Weekly for the duration of the study, approximately 15 weeks
  Subject's will walk at their self-selected speed while performing 1 of 4 cognitive tasks. Tasks include: serial subtraction, listing words in a specific category, reciting every other letter of the alphabet, repeating a list of numbers. The change in stride length and cadence were compared to baseline gait (walking at 3 speeds: normal, slow, fast) using the residual standard deviation (RSD) method. RSD evaluates gait variability while accounting for changes in velocity.
Prosthetic Single Limb Support | Weekly for the duration of the study, approximately 15 weeks
  Prosthesis users are reported to spend less time in single limb support on the prosthetic side due to a lack of stability. Improved stability with an MPK could increase prosthetic single limb support. The outcome will be measured over a range of walking speeds using an instrumented walkway.
Hip/knee/ankle joint angles | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  Joint angle range of motion and angle at critical instances will be measured using 3D motion capture to evaluate changes in gait kinematics while using each knee.
6-minute walk test | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  The 6-Min Walk Test is a functional walking test that is considered to be reflective of performance of activities of daily living. Participants will be instructed to walk as far as they can in 6 min along a wide, 30.5m (100 ft) corridor with sufficient additional space for unobstructed 180° turns at each end. Participants are free to pause at any time during the test; however, the time will continue to run. The distance walked during 6-Min Walk Test will be recorded to the nearest foot.
Berg Balance Scale | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  The Berg Balance Scale has high validity and reliability in assessing balance in prosthesis users. The Berg Balance Scale consists of 14 functional balance tasks scored from 0 to 4, with a max score of 56. It will be administered by a physical therapist experienced with the measure and working with lower-limb amputees.
Amputee Mobility Predictor | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  The Amputee Mobility Predictor is designed specifically for assessing amputees before or after receiving a prosthesis and the score can be used to assign Medicare Functional Class Level (K-Level, secondary outcome). The 20 tasks include assessments of balance and mobility (most tasks scored from 0-2, maximum score 47) and will be administered by a certified prosthetist. Although comparison between devices is not its primary intent, the Amputee Mobility Predictor has widespread use among practitioners and researchers, providing a consistent means to compare results between studies.

SECONDARY OUTCOMES:
Gait Velocity | Weekly for the duration of the study, approximately 15 weeks
  The maximum and normal self selected velocity will be evaluated for change in mobility with the MPK.
Dual-task cognitive performance | Weekly for the duration of the study, approximately 15 weeks
  The subject's performance on the cognitive dual-tasks evaluated at each session will be evaluated for change in performance. Tasks include: serial subtraction, listing words in a specific category, reciting every other letter of the alphabet, repeating a list of numbers. Tasks will be evaluated for rate of performance and accuracy.
Dual-task difficulty | Weekly for the duration of the study, approximately 15 weeks
  Subject's will rate their perceived difficulty of performing each dual-task on a 7-point Likert scale with 1 representing the perception of a task being very easy and 7 representing the perception of a very difficult task.
Step Width | Weekly for the duration of the study, approximately 15 weeks
  Prosthesis users are reported to walk with a wider step width due to a lack of stability. Step width will be measured over a range walking speeds to assess differences in lateral stability between the two knees.
Prosthetic limb double support | Weekly for the duration of the study, approximately 15 weeks
  Prosthesis user spend longer transitioning their weight to the prosthetic side during gait. Shorter prosthetic limb double support (early support) would signify increased confidence in transitioning weight to the prosthetic side. The prosthetic limb double support will be measured for a range of walking speeds using an instrumented walkway.
K-Level | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  The Medicare Functional Classification Level assigned by the Amputee Mobility Predictor.
Physiological Cost Index | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  Physiological Cost Index (PCI) is a measure of energy cost and can serve as a proxy measure of oxygen cost. Subject's heart rate will be measured manually before (resting heart rate) and within 30 s of completion of the 6-Minute Walk Test (exertion heart rate). PCI was calculated as the difference between the exertion heart rate and resting heart rate divided by the average walking speed (m/s) of the 6-minute Walk Test. A lower PCI value represents less energy cost during walking.
L-test | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  The L-Test assesses multiple aspects of mobility including sit-to-stand, level ground gait, and turns. On the signal to start, participants are instructed to rise from their chair, walk 3m to a marked spot, make a 90° right turn, walk 7m to a marked spot, turn 180°, return 7m, make a 90° left turn, walk 3m, return to chair, and take a seat. The assessment will be performed twice and the average time of the performances will be used for analysis.
Prosthesis Evaluation Questionnaire | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  The Prosthesis Evaluation Questionnaire (PEQ) evaluates different aspects of prosthetic use. Participants will complete the Mobility, Utility, and Well-Being subscales and the Satisfaction questions using the original 100-point visual scale. The adapted Mobility subscale will be evaluated rather than the original ambulation and transfer subscales.
Ground Reaction Forces | At baseline and end of each phase (5 weeks) for the duration of the study, approximately 15 weeks
  The ground reaction forces measured from force plates in the ground will be used to evaluate gait symmetry between the two knees.
Study specific preference scale | At the end of each phase after the first introduction of the MPK (5 weeks) for the duration of the study, approximately 15 weeks
  Subjects will be asked to rate their overall preference between the two knees on a visual analog scale ranging from -50 to +50. Negative scores represent preference for the subjects' own mechanical knee. Positive scores represent preference for the study MPK. Score near 0 represent neutral preference between the knees.

CONTACTS AND LOCATIONS:
Overall Officials: Dobrivoje Stokic, MD, DSc, Study Director — Methodist Rehabilitation Center

REFERENCES:
- [Result] Howard CL, Wallace C, Perry B, Stokic DS. The utility of the single-subject method for comparison of temporal-spatial gait changes between a microprocessor and non-microprocessor prosthetic knees. Prosthet Orthot Int. 2020 Jun;44(3):133-144. doi: 10.1177/0309364620909049. Epub 2020 Mar 18. PMID 32186241